CLINICAL TRIAL: NCT06016231
Title: Clinial Outcomes of Bilateral Pseudophakic Patients with a Light Adjustable Lens (LAL) Implanted in At Least One Eye
Brief Title: Clinical Outcomes of Patients with a Light Adjustable Lens (LAL) in At Least One Eye
Status: Completed | Type: Observational
Sponsor: Bucci Laser Vision Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-004
Record Dates: First submitted 2023-08-17; First posted 2023-08-29 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2023-08

CONDITIONS: IOL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- LAL in at least one eye
  Interventions: Device: Light Adjustable Lens

INTERVENTIONS:
Device: Light Adjustable Lens — The Light Adjustable Lens (LAL) is a posterior chamber, UV absorbing, three-piece, foldable, photoreactive silicone intraocular lens with a squared posterior optic edge intended to be implanted in the capsular bag following phacoemulsification. Selective exposure of the implanted RxSight LAL using the Light Delivery Device (LDD) to deliver a spatially profiled UV light produces modifications in the lens curvature resulting in a spherical or spherocylindrical power change post-operatively. A subsequent lock-in exposure is delivered to the implanted LAL to stabilize the lens power.

SUMMARY:
To collect data on bilateral pseudophakic patients implanted with the RxSight Light Adjustable Lens (LAL) in at least one eye

ELIGIBILITY:
Inclusion Criteria:

* Adults with bilateral pseudophakia who have been implanted with the LAL in at least one eye and who have completed LDD light treatments

Exclusion Criteria:

* Visually significant eye disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bilateral pseudophakia in adults implanted with the LAL in at least one eye and who have completed Light Delivery Device (LDD) light treatments
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction - subjective questionnaire | 3-18 months after cataract surgery
  Subjective questionnaire explores the frequency/need for glasses for various visual functions at distance/intermediate/near, experience with dysphotopsias, and overall satisfaction of visual function without glasses.

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Bucci, MD, Principal Investigator — Bucci Laser Vision Institute
Locations (1):
- Bucci Laser Vision Institute, Wilkes-Barre, Pennsylvania, United States